CLINICAL TRIAL: NCT05840848
Title: Effect of Simultaneously Consuming Iron and Zinc Supplements With That of B-carotene, on the B-carotene Bioavailability in Healthy Males
Brief Title: Effect of Iron and Zinc Supplementation on B-carotene Bioavailability in Healthy Males
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hohenheim (Other)
Responsible Party: Principal Investigator, Johanita Kruger, Dr. (PhD), University of Hohenheim
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: AZ: F-2017-039
Record Dates: First submitted 2023-03-28; First posted 2023-05-03 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Bioavailability
Keywords: B-carotene; Iron; zinc; Supplements
MeSH Terms: interventions — Iron-Dextran Complex

STUDY DESIGN:
Intervention Model Description: double-blind crossover
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control plus Placebo (Active Comparator): B-carotene supplement (15 mg) consumed in the morning after a >10 hour overnight fast.
  Interventions: Dietary Supplement: Control beta-carotene supplement plus Placebo
- Control plus iron Supplement (Experimental): B-carotene supplement (15 mg) and iron sulphate supplement (25 mg) consumed in the morning after a >10 hour overnight fast.
  Interventions: Dietary Supplement: Control beta-carotene supplement plus iron Supplement
- Control plus zinc Supplement (Experimental): B-carotene supplement (15 mg) and zinc sulphate supplement (30 mg) consumed in the morning after a >10 hour overnight fast.
  Interventions: Dietary Supplement: Control beta-carotene supplement plus zinc Supplement

INTERVENTIONS:
Dietary Supplement: Control beta-carotene supplement plus Placebo — 15 mg beta-carotene supplement from BIOVEA consumed before breakfast together with an empty capsule.
  Arms: Control plus Placebo
Dietary Supplement: Control beta-carotene supplement plus iron Supplement — 15 mg Beta-carotene supplement from BIOVEA consumed before breakfast together with 25 mg iron (FeSO4; Woerwag Pharma GmbH & Co. KG, Boeblingen, Germany)
  Arms: Control plus iron Supplement
Dietary Supplement: Control beta-carotene supplement plus zinc Supplement — 15 mg Beta-carotene supplement from BIOVEA consumed before breakfast together with 30 mg zinc (ZnSO4; Woerwag Pharma GmbH & Co. KG, Boeblingen, Germany)
  Arms: Control plus zinc Supplement

SUMMARY:
In vitro studies found supplemental levels of iron and zinc to inhibit the micellization and cellular uptake of β-carotene. Here, we investigated this in vivo, in a double-blind 3-arm crossover human trial.

Healthy males (n=6) ingested, with breakfast, a single dose of 15 mg β-carotene in combination with either a placebo, 25 mg iron or 30 mg zinc capsule. Blood samples were collected at baseline and hourly for 10 hours. The triacylglycerol-rich fraction (TRF) was analysed for concentrations of β-carotene and plasma for β-carotene, retinol, triacylglycerols, LDL- and HDL-cholesterol.

DETAILED DESCRIPTION:
The study followed a double-blind crossover design with three study arms separated by one week washout periods. In short, the participants were asked to follow a diet low in carotenoids by avoiding all orange, yellow, red and green fruits and vegetables for four days. This was followed by three days of a strictly carotenoid-free diet, which only allowed foods from a specified list (Supplemental Table A2). On each study day, β-carotene was administered in the morning after a >10 hour overnight fast (Supplemental Figure A1). All participants orally ingested, in random order, a single dose of 15 mg β-carotene (BIOVEA) with either a placebo (empty capsule), 25 mg iron (FeSO4; Woerwag Pharma GmbH & Co. KG, Boeblingen, Germany) or 30 mg zinc (ZnSO4; Woerwag Pharma) capsule. A standardised dinner was provided on the evening before the trial and standardised meals were provided during the entire intervention day (Supplemental Table A3). On the first study day, the amount of food (weight or volume) consumed by each participant for each meal was recorded and the same amounts provided during the following two arms to ensure similar food consumption, especially of fat. Water was available unrestricted for consumption throughout the day. Blood samples were drawn from an indwelling venous cannula and collected at 0 hours directly before β-carotene supplementation and then every hour for 10 hours.

For the determination of plasma concentrations of β-carotene, LDL- and HDL-cholesterol, and triacylglycerols (TAG), blood was collected in tubes containing EDTA (Sarstedt AG & Co, Nuebrecht, Germany) and immediately centrifuged (3000 × g, 10 min, 4 °C). From the obtained plasma samples, three aliquots were stored at -80 °C until further analysis and the rest ultracentrifuged to obtain the triacylglycerol-rich fraction (TRF). For the analyses of liver and kidney function markers, plasma and serum were obtained from blood sampled at the 0- and 4-hour time points.

The TRF was prepared according to [10]. Briefly, plasma (3.5 mL) was transferred to an ultracentrifuge tube and carefully overlaid with 8 mL 1.3% sodium chloride and then ultracentrifuged (Beckman Coulter, OptimaTM L-80 XP Ultracentrifuge) using a swinging bucket rotor (SW41Ti) at 150 000 x g for 1 hour at 4 °C. Afterwards, the TRF was isolated by transferring the upper ~6 mL, which was then overlaid with nitrogen gas to minimize oxidation and stored at -80 °C until extraction.

The plasma samples were randomly extracted and analysed by HPLC according to [15]. Briefly, 40 µL plasma was extracted with an ethanol/n-butanol mixture (50:50) containing apo-80-carotenal-methyloxime (12µL/100 mL; Fluka Analytical (Merck Group KGaA), Darmstadt, Germany) as internal standard. After centrifugation, the clear supernatant was analysed by HPLC.

The TRF was extracted and analysed by HPLC [15]. For the extraction, 100 µl apo-80-carotenal-methyloxime (12 µL/100 mL) and 2 mL ethanol (for deproteination) were added to 3 mL of the TRF and vortexed for 30 sec. The solution was extracted twice with 2 mL hexane. The hexane layers were removed, combined and evaporated in a centrifugal vacuum concentrator (Christ, RVC 2-25 CD plus) and the dried sample re-dissolved in 100 µL acetonitrile and immediately analysed by HPLC.

Both the plasma and TRF samples were analysed using a Shimadzu HPLC (LC-10AD) equipped with a UV-Vis detector (SPD 20A, set at 450 nm). Carotenoids were separated using a ReproSil 80 ODS-2 column (3 µm, 250 x 4.6 mm; Dr. Maisch GmbH, Ammerbuch, Germany) and an eluent in recirculation mode (82% acetonitrile, 15% 1,4-dioxin, and 3% methanol (vol/vol) containing 100 mM ammonium acetate and 10 mM triethylamine) at a flow rate of 1.5 mL/min [15]. A β-carotene standard (≥97.0% purity, Sigma-Aldrich) was used to construct a standard curve.

Plasma TAG, HDL- and LDL-cholesterol were analysed by a clinical laboratory (Laborärzte Sindelfingen, Sindelfingen, Germany).

ELIGIBILITY:
Inclusion Criteria:

* Male
* aged 18 and 50 years

Exclusion Criteria:

* overweight (BMI >25 kg/m2),
* metabolic and endocrine diseases,
* drug abuse,
* use of dietary supplements,
* us of any form of medication,
* smoking,
* frequent alcohol consumption (>20 g ethanol/day),
* adherence to a restrictive dietary regimen,
* physical activity of more than 5 h/wk,
* participation in a clinical trial within the past 3 months prior to recruitment,
* a known intolerance against β-carotene, iron and/or zinc supplements.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women were excluded from the study because the concentrations and distribution of carotenoids in the lipoprotein fractions fluctuate throughout the menstrual cycle
Enrollment: 12 (Actual)
Dates: Start 2017-11-21 (Actual); Primary Completion 2017-12-14 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
TRF B-carotene | 10 hours
  B-carotene concentration in the triacylglycerol-rich fraction of the plasma
Plasma B-carotene | 10 hours
  B-carotene concentration int he plasma

SECONDARY OUTCOMES:
Plasma LDL-cholesterol | 10 hours
  LDL-cholesterol concentration in Plasma
Plasma HDL-cholesterol | 10 hours
  HDL-cholesterol concentration in Plasma
Plasma TAG | 10 hours
  triacylglycerol concentration in Plasma
liver function markers | 4 hours
  γ-GT, AST, ALT, Alkaline phosphatase and Bilirubin measured
Kidney funtion markers | 4 hours
  Creatinine i.S. and Uric acid measured

CONTACTS AND LOCATIONS:
Locations (1):
- University of Hohenheim, Stuttgart, Baden-Wurttemberg, Germany

REFERENCES:
- [Derived] Kruger J, Sus N, Moser A, Scholz S, Adler G, Venturelli S, Frank J. Low beta-carotene bioaccessibility and bioavailability from high fat, dairy-based meal. Eur J Nutr. 2024 Sep;63(6):2261-2270. doi: 10.1007/s00394-024-03423-w. Epub 2024 May 16. PMID 38753174

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-10-02): https://cdn.clinicaltrials.gov/large-docs/48/NCT05840848/Prot_SAP_ICF_000.pdf